CLINICAL TRIAL: NCT04177017
Title: Learning Mindfulness Based Practices, Empathy and Pro-social Behavior in the Educational Field: Its Influence on Health and Interpersonal Relationships
Brief Title: Mindfulness, Empathy and Social Integration. Its Relation With Chonic Stress
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Council of Scientific and Technical Research, Argentina (Other Government)
Responsible Party: Principal Investigator, Paola D'Adamo, Researcher, National Council of Scientific and Technical Research, Argentina
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CONICET
Record Dates: First submitted 2019-11-22; First posted 2019-11-26 (Actual); Last update posted 2019-11-26 (Actual); Status verified 2019-11

CONDITIONS: Chronic Stress Disorder
Keywords: stress; empathy; sociality; cortisol
MeSH Terms: conditions — Social Behavior

STUDY DESIGN:
Intervention Model Description: semi-randmized controlled intervention
Masking Description: The lab that analyzed hair cortisol levels did not know to which group corresponded the samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): The experimental group is the one that participates in the intervention
  Interventions: Behavioral: Mindfulness-based intervention
- Control group (No Intervention): The control group belonged to the same school but did not participate in the intervention. Instead, they continued with regular curricular classes

INTERVENTIONS:
Behavioral: Mindfulness-based intervention — The behavioral intervention was carried out once a week during 60 minutes from May to November, and included mindfulness-based practices sought to foster self-awareness, and dyadic activities sought to awakening subtle perception of the other.
  Group activities, which entailed more than two participants, were also conducted to foster empathic collaboration and prosocialness. Diverse collaborative games were carried out in which mutual help was needed for achieving shared goals in an amusing way .
  Perspective-taking was encouraged within the group, by sharing each participant's experience, which included expressing how each child had felt (i.e., if neglected, ignored or cared for) and whether they had enjoyed helping their peers or no.
  Other Names: Self-awareness practices, and other oriented awareness practicess
  Arms: Experimental group

SUMMARY:
The objective of this project is to evaluate the effects of promoting the learning of empathy and pro-social behavior in health and interpersonal relationships in middle-aged children It has been shown that pro-social behavior can decrease chronic stress levels and improve the response of the immune system and the autonomic nervous system. This behavior, which includes a wide variety of actions such as helping, sharing, comforting, informing, emerges early in ontogeny and is closely related to empathic processes. Finding ways to teach how to develop empathy and perspective could contribute to favor interpersonal relationships and health in the school environment, articulating aspects of basic science and applied science. The project not only aims to deepen theoretical aspects of chornic stress, empathy and pro-sociality, but also to develop concrete tools that diminsh chronic stress and foster empathic and cooperative attitudes in the school environment, thus contributing to individual and collective well-being.

DETAILED DESCRIPTION:
The study will be carried out in primary educational establishments. In the experimental group, the proposed intervention will be conducted during the school year. The control group, with similar characteristics, will carry out regular curricular activities.

Informative talks will be given to parents of potential participants, teachers and managers of educational establishments, in order to inform about research objectives and methodology. The nature of voluntary participation in any of the activities and procedures, as well as the confidential treatment of the information will be duly clarified. Informed consent will be requested from parents if they agree to participate in the project.

The intervention program will consist of a weekly meeting of approximately 1 hour during the school year, and will be conducted by the researchers together with the teacher in charge of the group. This program will include practices that promote self-perception, interoception and collaborative activities, followed by an instance of group reflection that promotes perspective taking (as in Lozada et al 2017).

The practices of self-perception and interoception consist, for example, in focusing attention on breathing for a period of time that will gradually increase (mindfulness). During collaborative actions, children will carry out activities in dyads or in small groups that promote empathy and pro-social behavior. The last activity of the intervention will consist of an instance of group reflection in which experiences and perceptions of the participants will be shared in order to favor perspective taking (i.e. the cognitive ability to consider the world from the point of view of the other).

The variables (pro-social behavior and hair cortisol levels) are quantified at the beginning and at the end of each intervention (ie, pre and post-test evaluation). To assess the differences in each group, pre-post levels will be compared by means of the paired t test, and comparisons between the experimental and control groups will be made by means of variance analysis tests and Mann Withney tests and Kruskal Wallis.

Children participating in the experimental and control groups will be individually evaluated using the following methods:

3) Sociometric questionnaire.

Stress levels are quantified through:

1) Hair cortisol dosing. This parameter is an indicator of chronic stress whose advantage is that it does not show marked variability throughout the day such as salivary cortisol. For this, it is necessary to cut a small strand of hair that will be analyzed later by Pharmacy and Biochemistry researchers from the University of Buenos Aires.

ELIGIBILITY:
Inclusion Criteria:

* Participants having good general health

Exclusion Criteria:

* Children who were taking medication
* Children that were present to less than the 80% of the intervention encounters
* Children who were not present at the pre and post measurements points

Ages: 6 Years to 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 35 (Actual)
Dates: Start 2017-03-20 (Actual); Primary Completion 2017-11-30 (Actual); Study Completion 2018-06-23 (Actual)

PRIMARY OUTCOMES:
Change from baseline hair cortisol levels | through study completion, an average of 9 months
  change form baseline hair cortisol levels at 9 months
change from baseline sociogram levels | through study completion, an average of 9 months
  Children are asked to say which classmates they would choose as playmates and which ones they would not. The sociogram is completed previous to and after the intervention in both groups. The changes in the number of peers selected (i.e., positive elections) and rejected (i.e., negative elections) reflect changes in the pattern of social relationships of each child. Therefore, if positive elections increase and /or negative elections decrease, social integration improves

CONTACTS AND LOCATIONS:
Overall Officials: Paola D'Adamo, PhD, Principal Investigator — National Council of Scientific and Technical Research, Argentina
Locations (1):
- Paola, Bariloche, Río Negro Province, Argentina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Iglesias S, Jacobsen D, Gonzalez D, Azzara S, Repetto EM, Jamardo J, Gomez SG, Mesch V, Berg G, Fabre B. Hair cortisol: A new tool for evaluating stress in programs of stress management. Life Sci. 2015 Nov 15;141:188-92. doi: 10.1016/j.lfs.2015.10.006. Epub 2015 Oct 22. PMID 26454227
- [Result] Lozada M, Carro N, D'adamo P, Barclay C. Stress management in children: a pilot study in 7 to 9 year olds. J Dev Behav Pediatr. 2014 Feb-Mar;35(2):144-7. doi: 10.1097/DBP.0000000000000026. PMID 24406660